CLINICAL TRIAL: NCT02862860
Title: Influence of Glycaemic Variability on Oxidative Stress and High-density Lipoprotein (HDL) Function in Type-1 Diabetes
Brief Title: Search for a Link Between the Different Variables for Glycaemia and Oxidative Stress or Impaired HDL Function
Acronym: Holter Gly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: Duvillard Hors AOI 2011
Record Dates: First submitted 2016-07-28; First posted 2016-08-11 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Type-1 Diabetes
MeSH Terms: interventions — Blood Specimen Collection

ARMS (2):
- patients with type-1 diabetes (Experimental)
  Interventions: Biological: blood sample; Biological: urine sample; Device: installation of Holter
- Controls (Placebo Comparator)
  Interventions: Biological: blood sample; Biological: urine sample

INTERVENTIONS:
Biological: blood sample
Biological: urine sample
Device: installation of Holter
  Arms: patients with type-1 diabetes

SUMMARY:
As glycaemic variability on the one hand and hypoglycaemia on the other are associated with oxidative stress and inflammation, they are likely, in type-1 diabetic patients, to affect the oxidation of lipoproteins and HDL function, by altering their anti-atherogenic properties.

The aim of this study is thus to determine, in patients with Type 1 Diabetic (T1D) who will wear a glycaemic Holter for 1 week, the glycaemia parameters (mean glycaemia, duration of hypoglycaemia, duration of hyperglycaemia, mean amplitude of glycaemic excursions) associated with proatherogenic alterations in lipoproteins, in particular:

* LDL oxidation
* HDL oxidation and alterations of HDL function (anti-inflammatory capacity, antioxidant capacity)

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided written consent
* Patients with national health insurance cover

Patients with T1D

* T1D Patients treated with insulin via a pump or multiple injections
* HbA1c < 9.5 %

Control patients

* Normal fasting glycaemia (< 6.1 mmol/L)
* Age > 18 years, matched for sex and age with T1D patients

All patients

* Normal serum HDL cholesterol (> 1.04 mmol/L in men, > 1.30 mmol:L in women)
* Serum LDL cholesterol < 5 mmol/L
* triglyceridemia < 1.7 mmol/L
* Waist circumference < 102 cm in men, < 88 cm in women

Exclusion Criteria:

* Smoking
* Kidney failure (Creatinine clearance< 60 ml/min/1.73 m2)
* Liver failure
* Dysthyroidism
* Medication that interferes with lipoprotein metabolism (lipid-lowering agents, oestroprogestative, anti-HIV, corticoids, retinoic acid), unless stopped for at least one 1 month
* Antioxidant (vitamin E, dietary supplements, DHA)
* Pregnancy of more than 15d

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-05-29 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2018-04-17 (Actual)

PRIMARY OUTCOMES:
Average blood glucose | through study completion, an average of 7 days
Time hypoglycemia | through study completion, an average of 7 days
Time hyperglycemia | through study completion, an average of 7 days
Amplitude of glycemic variations | through study completion, an average of 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France